CLINICAL TRIAL: NCT04534517
Title: Clinical Evaluation of a Daily Wear Reusable Multifocal Optical Design in a Presbyopic Population
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Vision Care, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR-6400
Record Dates: First submitted 2020-08-27; First posted 2020-09-01 (Actual); Results first posted 2022-01-13 (Actual); Last update posted 2022-01-13 (Actual); Status verified 2021-12

CONDITIONS: Visual Acuity

STUDY DESIGN:
Masking Description: Participant is masked to the brand of the devices
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- TEST Lens (Experimental): Eligible subjects who are habitual soft contact lens wearers between the ages of 40 and 70 years of age will be recruited. Alternative Spherical lenses will be used if optimization cannot be achieved with the Multifocal lenses.
  Interventions: Device: JJV Investigational Multifocal Contact Lens; Device: ACUVUE OASYS® with HYDRACLEAR® PLUS

INTERVENTIONS:
Device: JJV Investigational Multifocal Contact Lens — TEST Lens
Device: ACUVUE OASYS® with HYDRACLEAR® PLUS — The spherical test lens was used in the troubleshooting steps only for low ADD subjects who have reported a distance vision complaint.
  Other Names: senofilcon A

SUMMARY:
The clinical study is a bilateral, single-masked (partial), single-arm, clinical trial. A total of approximately 60 eligible subjects both near-sighted and far-sighted, will be targeted to complete the study. Subjects will be fit in the study lens for approximately 2-4 days then undergo lens optimization, if required. Subjects will then be given a new pair of lenses that will be worn for approximately 2 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. The subject must read, understand, and sign the STATEMENT OF INFORMED CONSENT and receive a fully executed copy of the form.
2. The subject must appear able and willing to adhere to the instructions set forth in this clinical protocol.
3. The subject must be at least 40 years of age and not greater than 70 years of age at the time of consent.
4. Subjects must own a wearable pair of spectacles if required for their distance vision.
5. The subject must be an adapted soft contact lens wearer in both eyes (i.e. wears lenses a minimum of 2 days per week for at least 6 hours per wear day, for 1 month of more duration).
6. The subject must either already be wearing a presbyopic contact lens correction (e.g., reading spectacles over contact lenses, multifocal or monovision contact lenses, etc.) or if not respond positively to at least one symptom on the "Presbyopic Symptoms Questionnaire" (Appendix E).
7. The subject's distance spherical equivalent refraction (vertex corrected if ≥-4.25 D) must be in the range of -1.25 D to -5.75 D or +0.75 D to +3.25 D in each eye.
8. The subject's refractive cylinder must be ≤0.75 D in each eye.
9. The subject's ADD power must be in the range of +0.75 D to +2.50 D.
10. The subject must have distance best corrected visual acuity of 20/20-3 or better in each eye.

Exclusion Criteria:

1. Currently pregnant or lactating.
2. Any active or ongoing ocular or systemic allergies that may interfere with contact lens wear.
3. Any active or ongoing systemic disease, autoimmune disease, or use of medication, which may interfere with contact lens wear. This may include, but not be limited to, diabetes, hyperthyroidism, Sjögren's syndrome, xerophthalmia, acne rosacea, Stevens-Johnson syndrome, and immunosuppressive diseases or any infectious diseases (e.g. hepatitis, tuberculosis).
4. Any previous, or planned, ocular or intraocular surgery (e.g. radial keratotomy, PRK, LASIK, lid procedures, dacryocystorhinostomy, peripheral iridotomy/iridectomy, cataract surgery, retinal surgery, etc.).
5. A history of amblyopia, strabismus or binocular vision abnormality.
6. History of glaucoma, macular degeneration, recurrent corneal erosions, recurrent styes, herpetic keratitis, irregular cornea or pathological dry eye.
7. Use of any of the following medications within 1 week prior to enrollment: oral retinoids, oral tetracyclines, oral phenothiazines, anticholinergics, corticosteroids.
8. Use of any ocular medication, with the exception of rewetting drops.
9. Participation in any contact lens or lens care product clinical trial within 30 days prior to study enrollment.
10. Employee or immediate family member of an employee of clinical site (e.g., Investigator, Coordinator, Technician).
11. Any known hypersensitivity or allergic reaction to Optifree® Replenish® multipurpose care solution, sodium fluorescein or non-preserved rewetting drop solutions.
12. Clinically significant (Grade 2 or greater) corneal edema, corneal vascularization, corneal staining, tarsal abnormalities or bulbar injection, or any other corneal or ocular abnormalities which would contraindicate contact lens wear.
13. Any current ocular infection or inflammation.
14. Any current ocular abnormality that may interfere with contact lens wear.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 119 (Actual)
Dates: Start 2020-08-07 (Actual); Primary Completion 2020-09-29 (Actual); Study Completion 2020-09-29 (Actual)

CONTACTS AND LOCATIONS:
Locations (11):
- United States (11):
  - Dr. James Weber & Associates, PA, Jacksonville, Florida
  - Sabal Eye Care, Longwood, Florida
  - Maitland Vision Center, Maitland, Florida
  - VisualEyes, Roswell, Georgia
  - VisionPoint Eye Center, Bloomington, Illinois
  - Kannarr Eye Care, Pittsburg, Kansas
  - Advanced Eyecare, Raytown, Missouri
  - Sacco Eye Group, Vestal, New York
  - ProCare Vision Centers, Granville, Ohio
  - Dr. David W. Ferris & Associates, Warwick, Rhode Island
  - Frazier Vision Inc., Tyler, Texas

IPD SHARING:
Plan to Share IPD: Yes
Johnson & Johnson Medical Device Companies have an agreement with the Yale Open Data Access (YODA) to serve as the independent review panel for evaluation of requests for clinical study reports and participant level data from investigators and physicians for scientific research that will advance medical knowledge and public health. Requests for access to the study data can be submitted through the YODA Project site at http://yoda.yale.edu
URL: http://yoda.yale.edu

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 119 subjects were enrolled into this study. Of those enrolled, 114 subjects were dispensed a study lens while 4 subjects failed to meet all eligibility criteria. Of those dispensed, 110 completed the study while 4 subjects were discontinued.
Groups:
- Senofilcon A (Investigational Multifocal Lens): All subjects that wore the investigational multifocal lens made from senofilcon A material during the entire duration of the study.
Period: Overall Study
Arm/Group | Senofilcon A (Investigational Multifocal Lens)
Started | 114
Completed | 110
Not Completed | 4
Not completed — Adverse Event | 1
Not completed — Withdrawal by Subject | 1
Not completed — Unsatisfactory Visual Response due to Test Article | 1
Not completed — COVID-19 Related | 1

BASELINE CHARACTERISTICS:
Groups:
- Hyperopes; Myopes: All subjects dispensed a study lens.
- Total: Total of all reporting groups
Arm/Group | Hyperopes | Myopes | Total
Number analyzed (Participants) | 55 | 59 | 114
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.8 (6.78) | 50.5 (6.21) | 53.5 (7.21)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 49 | 48 | 97
  Male | 6 | 11 | 17
Race/Ethnicity, Customized [Number; unit: participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Black or African American | 3 | 3 | 6
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  White | 50 | 56 | 106
Region of Enrollment [Number; unit: participants]
  United States | 55 | 59 | 114

OUTCOME MEASURES:

1. Primary Outcome: Vision Scores
Description: Overall vision scores were assessed using the Contact Lens User Experience™ (CLUE) questionnaire. CLUE is a validated patient-reported outcomes (PRO) questionnaire to assess patient experience attributes of soft contact lenses (comfort, vision, handling, and packaging) in a contact-lens wearing population in the US, ages 18-65. Derived CLUE scores using Item Response Theory (IRT) follow a normal distribution with a population average score of 60 (SD 20), where higher scores indicate a more favorable/positive response with a range of 0-120. The average CLUE vision score for each sphere stratum (Hyperope and Myope) was reported.
Time Frame: 2-Week Follow-up
Population: All subjects that completed all study visits without a major protocol deviation impacting a primary endpoint.
Measure: Mean (Standard Deviation); unit: CLUE points
Arm/Group | Senofilcon A (Investigational Multifocal Lens)
Number analyzed (Participants) | 105
CLUE points
  Hyperopes: number analyzed (Participants) | 50
  Hyperopes | 57.48 (21.175)
  Myopes: number analyzed (Participants) | 55
  Myopes | 61.97 (20.671)
Statistical Analysis 1: Comparison: Senofilcon A (Investigational Multifocal Lens); It was calculated that 60 participants would have > 99% power to for the mean CLUE vision scores for each sphere stratum to be above the hypothesis threshold at the 2-week follow-up. Sample size was determined using one sample means test for equivalence; Test type: Superiority — The superiority of the Test lens was concluded if the lower credible limit of the mean was above the pre-defined threshold 32 points; Bayesian multivariate random-effects; Mean Estimate = 58.6, 95% CI 2-sided [52.3 to 64.9], Standard Deviation 3.26 — Included Hyperope group only
Statistical Analysis 2: Comparison: Senofilcon A (Investigational Multifocal Lens); [analysis description as in outcome 1, analysis 1]; Test type: Superiority — The superiority of the Test lens was concluded if the lower credible limit of the mean was above the pre-defined threshold 40 points for Myopes; Bayesian multivariate random-effects; Mean Estimate = 63.8, 95% CI 2-sided [57.9 to 69.6], Standard Deviation 2.97 — Included myope group only

2. Primary Outcome: Visual Performance LogMAR
Description: Binocular visual performance on logMAR (Logarithm of Minimal Angle of Resolution) scale was evaluated at distance (4m), intermediate (64cm) and near (40cm) under high luminance high contrast lighting condition using ETDRS (Early Treatment Diabetic Retinopathy Study) charts. The room illuminance was required to be between 7.3 to 7.9 EV (394-597 lux). For Distance (4m), the acceptable range for the chart luminance was 10.5-10.7 EV (181 208 cd/m2). For Intermediate (64cm) and Near (40cm), the acceptable range for the chart luminance 10.8-11.1 EV (223-274 cd/m2). Letter-by-letter results calculated the visual performance score for each chart read. A logMAR score closer to zero, or below zero, indicates a better visual acuity. A logMAR visual performance score of 0.0 is equivalent to Snellen visual acuity of 20/20. Data from hyperopes and myopes were combined for this outcome since logMAR scores between the two populations are similar.
Time Frame: 2-Week Follow-up
Population: All subjects that completed all study visits without a major protocol deviation impacting a primary endpoint. Hyperopes and myopes were combined based on historical data for subjects in this study with regard to visual performance logMAR.
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | Senofilcon A (Investigational Multifocal Lens)
Number analyzed (Participants) | 105
logMAR
  Distance (4M) | -0.09 (0.105)
  Intermediate (64 cm) | -0.06 (0.084)
  Near (40 cm) | 0.06 (0.086)
Statistical Analysis 1: Comparison: Senofilcon A (Investigational Multifocal Lens); It was calculated that 60 participants would have > 99% power to for the mean visual performance at each distance to be below the hypothesis threshold at the 2-week follow-up. Sample size was determined using one sample means test for equivalence; Test type: Superiority — The superiority of the Test lens was concluded if the upper credible limit of the mean was below the pre-defined threshold +0.10 logMAR for Distance; Bayesian normal random-effects model; Repeated Measures; Mean estimate = -0.090, 95% CI 2-sided [-0.125 to -0.057], Standard Deviation 0.0172
Statistical Analysis 2: Comparison: Senofilcon A (Investigational Multifocal Lens); [analysis description as in outcome 2, analysis 1]; Test type: Superiority — The superiority of the Test lens was concluded if the upper credible limit of the mean was below the pre-defined threshold +0.17 logMAR for Intermediate; Bayesian normal random-effects model; Repeated Measures; Mean Estimate = -0.057, 95% CI 2-sided [-0.091 to -0.024], Standard Deviation 0.0171
Statistical Analysis 3: Comparison: Senofilcon A (Investigational Multifocal Lens); [analysis description as in outcome 2, analysis 1]; Test type: Superiority — The superiority of the Test lens was concluded if the upper credible limit of the mean was below the pre-defined threshold +0.17 logMAR for Near; Bayesian normal random-effects model; Repeated Measures; Mean Estimate = 0.066, 95% CI 2-sided [0.031 to 0.098], Standard Deviation 0.0171

3. Primary Outcome: Proportion of Eyes With Unacceptable Lens Fitting
Description: Contact lens fitting acceptance was assessed for each subject eye using a biomicroscope post lens insertion and the 2-week follow-up. Lens fit was a binary variable where acceptable lens fit=1 and unacceptable lens fit=0. The proportion of eyes with unacceptable lens fit was reported. Data from the hyperope and myopes group were combined for this outcome since lens fitting characteristerics are similar for these two populations.
Time Frame: Up to 2-Week Follow-up
Population: All subjects were dispensed at least one study lens.
Measure: Number; unit: proportion of eyes
Units Other Than Participants: Eyes
Arm/Group | Senofilcon A (Investigational Multifocal Lens)
Number analyzed (Participants) | 114
Number analyzed (Eyes) | 228
proportion of eyes | 0
Statistical Analysis 1: Comparison: Senofilcon A (Investigational Multifocal Lens); Test type: Superiority — A superiority margin of 5% was used. Upper limit of 95% credible interval was compared to 5%; Bayesian beta-binomial model; Correlated Binary Data; Mean Proportion = 0.001, 95% CI 2-sided [0.000 to 0.004], Standard Deviation 0.0012

4. Primary Outcome: Proportion of Eyes With Grade 3 or Higher Slit Lamp Findings
Description: Slit Lamp Findings (SLF) were assessed using a biomicroscope and was graded using the FDA grading scale (Grade: 0, 1,2, 3 and 4) with grade 0 represents the absence of findings and 1 to 4 representing successively worse findings (i.e. Grade 1 = trace, Grade 2 = Mild, Grade 3 = moderate and Grade 4 = severe). This was performed on each subject eye at every study visit (baseline, unscheduled visits and 2-week follow-up). The data was then dichotomized into two groups. Those with grade 3 or higher and those with grade 2 or lower. The proportion of eyes with SLF with grade 3 or higher was reported. Data from the hyperope and myopes group were combined for this outcome since the rate of SLFs grade 3 + is similar for both populations.
Time Frame: Up to 2-Week Follow-up
Population: All subjects were dispensed at least one study lens.
Measure: Number; unit: proportion of eyes
Units Other Than Participants: Eyes
Arm/Group | Senofilcon A (Investigational Multifocal Lens)
Number analyzed (Participants) | 114
Number analyzed (Eyes) | 228
proportion of eyes | 0
Statistical Analysis 1: Comparison: Senofilcon A (Investigational Multifocal Lens); Test type: Superiority — A superiority margin of 5% was used. Upper limit of the 95% credible interval was compared to 5%; Bayesian beta-binomial model; Correlated Binary Data; Mean Proportion = 0.005, 95% CI 2-sided [0.000 to 0.018], Standard Deviation 0.0048

5. Secondary Outcome: Proportion of Eyes That Achieved Optimal Lens Pair in 4 Lenses or Less
Description: The number of lenses to achieve the optimal pair for each subject was calculated as the original pair (2) plus all the required modifications to reach the optimal pair. In this study the minimum number of lenses per subject used was 2 where the maximum possible number of lenses used was 12. The data was dichotomized as Y=1 if the subject was able to achieve optimal lens pair in 4 lenses or lenses or less and 0 otherwise. A lens modification was performed if the subject reports unsatisfactory vision or was unable to obtain 20/30 distance visual acuity in both eyes. If the subject reported satisfactory vision with the lenses a modification was not required. However, based upon the investigator's findings on the measured visual acuity and/or over-refraction a modification may have been performed. Data for the hyperope and myope groups were combined for this endpoint since the number of lenses needed to optimize vision is indpendent of which group a subject belongs to.
Time Frame: Up to 2-Week Follow-up
Population: All subjects were dispensed at least one study lens.
Measure: Number; unit: proportion of eyes
Units Other Than Participants: Eyes
Arm/Group | Senofilcon A (Investigational Multifocal Lens)
Number analyzed (Participants) | 114
Number analyzed (Eyes) | 228
proportion of eyes | 0.4
Statistical Analysis 1: Comparison: Senofilcon A (Investigational Multifocal Lens); Test type: Superiority — A superiority margin of 90% was used. Lower limit of the 95% credible interval was compared to 90%; Bayesian beta-binomial model; Correlated Binary Data; Mean Proportion = 0.992, 95% CI 2-sided [0.973 to 0.999], Standard Deviation 0.0072

ADVERSE EVENTS:
Time Frame: Throughout the duration of the study. Approximately 2 weeks per subject.
Arm/Group | Senofilcon A (Investigational Multifocal Lens)
All-Cause Mortality (participants affected / at risk) | 0/114
Serious Adverse Events (participants affected / at risk) | 0/114
Other Adverse Events (participants affected / at risk) | 0/114

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2020-08-06): https://cdn.clinicaltrials.gov/large-docs/17/NCT04534517/Prot_002.pdf
  • Statistical Analysis Plan (2020-11-03): https://cdn.clinicaltrials.gov/large-docs/17/NCT04534517/SAP_001.pdf